CLINICAL TRIAL: NCT00523926
Title: An Open-label Study to Evaluate the Extended Early Bactericidal Activity, Safety, Tolerability and Pharmacokinetics of Multiple Oral Doses of TMC207 in Treatment-na�ve Subjects With Sputum Smear Positive Pulmonary Tuberculosis.
Brief Title: TMC207-C202: Study to Evaluate Bactericidal Activity of Multiple Oral Doses of TMC207 in Subjects With Sputum-Smear Positive Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002725
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Tuberculosis
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — bedaquiline

INTERVENTIONS:
Drug: TMC207

SUMMARY:
The purpose of this study is to assess the effects of 3 different oral doses of TMC207 administered over a 7 day period on the organism that causes tuberculosis

DETAILED DESCRIPTION:
This is a Phase IIa, open-label, randomized trial in treatment-naïve, sputum smear-positive, subjects with pulmonary TB to assess the extended early bactericidal activity (eEBA) of TMC207. The study population will consist of 60 treatment-naive subjects with M. tuberculosis infection.

Subjects will receive orally 25 mg TMC207 po q.d. (Treatment A), 100 mg TMC207 po q.d. (Treatment B) or 400 mg TMC207 po q.d. (Treatment C) daily for 7 days. Subjects in treatment group D will receive 600 mg rifampin po q.d. daily for 7 days and subjects in treatment group E will receive 300 mg isoniazid po q.d. daily for 7 days. After 7 days, subjects in all treatment groups will receive appropriate anti-TB therapy according to national standards of country TB guidelines and culture and sensitivity results of the sputum specimens until clinical and microbiological cures have been achieved. Three once-daily dose regimens of TMC207, for 7 days, will be studied versus 2 comparator treatments, rifampin and isoniazid in the present trial.TMC207 treatment groups: 25 mg TMC207 po q.d; 100 mg. TMC207 po q.d; 400 mg TMC207 po q.d.; TMC207 will be administered as a 10 or 40 mg/mL oral solution. Comparator groups: 600 mg rifampin po q.d. administered as capsules containing 300 mg rifampin; 300 mg isoniazid po q.d. administered as tablets containing 300 mg isoniazid.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive subjects with pulmonary M. tuberculosis infection, willing to start anti-TB therapy
* Positive for acid-fast bacilli on direct smear exam of sputum specimen
* Must consent to HIV testing
* Must agree to hospital admission

Exclusion Criteria:

* History or presence of hepatic or GI disease that may interfere with the absorption of TMC207, isoniazid or rifampin
* Subjects who received previous anti-mycobacterial drugs for the treatment of a mycobacteria infection and subjects who have received more than 2 weeks of treatment with a fluoroquinolone
* Subjects who have received antiretroviral therapy and/or oral or I.V. anti-fungal medication w/in the last 90 days
* Subjects with sputum cultures of M. tuberculosis resistant to rifampin
* Impaired hepatic function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-05; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Assess the effects of 3 doses of TMC207 administered over a 7 day period on M. tuberculosis in sputum compared to effects of treatment with standard doses of isoniazid and rifampin

SECONDARY OUTCOMES:
Assess the short term safety, tolerability and PK of multiple oral doses of TMC207 in treatment-naïve subjects with pulmonary M.tuberculosis infection

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA

REFERENCES:
- [Result] Rustomjee R, Diacon AH, Allen J, Venter A, Reddy C, Patientia RF, Mthiyane TC, De Marez T, van Heeswijk R, Kerstens R, Koul A, De Beule K, Donald PR, McNeeley DF. Early bactericidal activity and pharmacokinetics of the diarylquinoline TMC207 in treatment of pulmonary tuberculosis. Antimicrob Agents Chemother. 2008 Aug;52(8):2831-5. doi: 10.1128/AAC.01204-07. Epub 2008 May 27. PMID 18505852